CLINICAL TRIAL: NCT05064111
Title: Improved Detection and Localization Accuracy of Early Aggressive Prostate Adenocarcinoma Using Novel MR-directed Ultrasound-guided (MRdUSg) Prostate Biopsy Technique
Brief Title: Utility of Adding MR Fusion to Standard US Guided Prostate Biopsy
Status: Suspended | Type: Observational
Why Stopped: Per PI, the project start is on suspension.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 2012285076
Record Dates: First submitted 2021-08-02; First posted 2021-10-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All subjects: The experimental conditions will include a standard prostate biopsy using an FDA-approved ultrasound machine with application of the experimental (non-FDA approved) image fusion software.
  Interventions: Diagnostic Test: TRUS biopsy

INTERVENTIONS:
Diagnostic Test: TRUS biopsy — The biopsy procedure will be completed using an FDA-approved ultrasound machine with the addition of an investigational (non-FDA approved) image fusion software.

SUMMARY:
The purpose of this study is to utilize this technology in the early detection and staging of pathologic states within prostate cancer patients using the information obtained on mpMRI and serum biomarkers from the patient's blood (if collected). Ultimately, investigators hope to improve the diagnostic accuracy and treatment selection process for these patients. Applying the fusion software which adds mpMRI to ultrasound images in real time, to an otherwise clinically standard but non-targeted ultrasound-guided prostate biopsy procedure will help with accurate and early diagnosis of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent
2. Male - age > 18
3. mpMRI within the previous 6 months (PIRADS 3,4,5, all stages of PCa)
4. Scheduled for TRUS biopsy for prostate lesion or mass

Exclusion Criteria:

1. Age under 18 years of age.
2. Female
3. Pre-existing blood dyscrasias
4. Inability to perform TRUS due to anal sphincter closure/surgery
5. Patients needing general anesthesia
6. Patients allergic to lidocaine
7. Patients allergic or unable to take antibiotics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male patients undergoing diagnostic work up for suspected or recurrent prostate cancer as standard of care.
Study Population: Adult male patients undergoing diagnostic work up for suspected or recurrent prostate cancer as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate investigational fusion software. | Through study completion, planned 5 year duration.
  To evaluate the sensitivity of the investigational software to aid in targeted biopsy of prostate lesions seen on pre-biopsy mpMRI.

SECONDARY OUTCOMES:
Assess accuracy of mpMRI. | Through study completion, planned 5 year duration.
  To assess the diagnostic accuracy of Multiparametric Magnetic Resonance Imaging (mpMRI) provided Prostate Imaging Reporting and Data System (PIRADS) with pathology as the reference standard. The research-only procedure of collecting blood will be drawn during the scheduled biopsy visit, using no more than 15 minutes when the subject would already be at the visit. TRUS biopsy is standard of care. Experimental software will be added during the TRUS biopsy, at the time of needle localization. The software performs a computation on the ultrasound machine that fuses the pre-biopsy mpMRI images with the real-time ultrasound images.
Assess sensitivity of software. | Through study completion, planned 5 year duration.
  To assess the sensitivity of the investigation software in successfully targeting clinically significant prostate cancer, defined as Gleason score of 3+4 or greater. The research-only procedure of collecting blood will be drawn during the scheduled biopsy visit, using no more than 15 minutes when the subject would already be at the visit. TRUS biopsy is standard of care. Experimental software will be added during the TRUS biopsy, at the time of needle localization. The software performs a computation on the ultrasound machine that fuses the pre-biopsy mpMRI images with the real-time ultrasound images.
Correlation of imaging with biomarkers. | Through study completion, planned 5 year duration.
  To correlate Prostate Imaging Reporting and Data System (PIRADS) score from Multiparametric Magnetic Resonance Imaging (mpMRI) with cellular/ molecular biomarkers of aggressive cancer in the biopsy tissue samples. The research-only procedure of collecting blood will be drawn during the scheduled biopsy visit, using no more than 15 minutes when the subject would already be at the visit. TRUS biopsy is standard of care. Experimental software will be added during the TRUS biopsy, at the time of needle localization. The software performs a computation on the ultrasound machine that fuses the pre-biopsy mpMRI images with the real-time ultrasound images.

CONTACTS AND LOCATIONS:
Overall Officials: Hina Arif-Tiwari, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States